CLINICAL TRIAL: NCT02281487
Title: Hysterectomy for Benign Gynaecological Conditions With or Without Tubectomy
Acronym: HYSTUB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynaecologisch Oncologisch Centrum Zuid (Other)
Collaborators: Elisabeth-TweeSteden Ziekenhuis (Other); Catharina Ziekenhuis Eindhoven (Other); Radboud University Medical Center (Other); Jeroen Bosch Ziekenhuis (Other)
Responsible Party: Principal Investigator, Jurgen M.J. Piek, MD. PhD., Gynaecologisch Oncologisch Centrum Zuid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HYSTUB; NL39317.028.12 (Other: CCMO)
Record Dates: First submitted 2014-07-01; First posted 2014-11-03 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Abdominal Hysterectomy (& Wertheim)
Keywords: tubal carcinoma; ovarian carcinoma; tubectomy; hysterectomy; dysplastic changes; Anti Mullerian Hormone; Tubal Intraepithelial Carcinoma; Salpingectomy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Hysterectomy; Salpingectomy; Microscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hysterectomy (Active Comparator): standard hysterectomy
  Interventions: Procedure: Hysterectomy
- Hysterectomy plus tubectomy (Experimental): Hysterectomy plus tubectomy
  Interventions: Procedure: Hysterectomy plus Tubectomy; Device: light microscopy

INTERVENTIONS:
Procedure: Hysterectomy plus Tubectomy — hysterectomy with tubectomy
  Arms: Hysterectomy plus tubectomy
Procedure: Hysterectomy — standard hysterectomy
  Arms: Hysterectomy
Device: light microscopy — analysis of the incidence of dysplastic lesions (defined as: nuclear atypia, pilling of epithelial cells, multiple mitosis), if any, in the removed Fallopian tubes by light microscopy (Leica DM4000)
  Arms: Hysterectomy plus tubectomy

SUMMARY:
The purpose of this study is to determine whether a tubectomy during hysterectomy for benign gynaecological conditions does not result into a premature menopause.

DETAILED DESCRIPTION:
RATIONALE Recent studies in women at hereditary high risk to develop ovarian cancer indicate that high grade serous carcinomas arise from (ectopic and/or dysplastic) tubal epithelium. Historically, in pre-menopausal women undergoing a hysterectomy for benign indications (such as bleeding disorders, fibroids and adenomyosis) adnexa, including the Fallopian tubes, are left in situ. However, removing the tubes during a hysterectomy potentially prevents the development of serous ovarian carcinomas. Such a simple preventive procedure should avoid serious adverse effects of adnexectomy, like premature ovarian failure (POF).

STUDY DESIGN This is a randomized controlled trial in which patients undergoing a hysterectomy for benign indications will either be included into a group in which a standard hysterectomy (abdominal or laparoscopic) will be performed or into a group in which hysterectomy (abdominal or laparoscopic) will be combined with salpingectomy.The accrual is aimed to take until July 2015 and will be performed in the regular clinical setting.

STUDY POPULATION Women undergoing hysterectomy for benign conditions (fibroids, endosalpingiosis, bleeding disorders, etc) either abdominal or laparoscopic.

SAMPLE SIZE N=50/arm

TREATMENT Hysterectomy (abdominal or laparoscopic) with or without bilateral tubectomy.

METHODS

1. Study endpoint Main study endpoint: serum concentration Anti Mullerian Hormone (AMH) just before the operation and on average six months after the operation.

   Secondary study endpoint: premalignant changes within the removed Fallopian tubes from this cohort of women, defined as histological dysplastic areas detected by light microscope
2. Randomization Randomization is performed online with Alea software.
3. Study procedures One day preoperative, together with regular blood drawing, blood for AMH concentration assessment is drawn. The operation procedure will either be the regular procedure or the regular procedure plus removal of the Fallopian tubes by removing the tubes from the ovaries by dissection of the mesovarium. On an expected average of six months after the operation blood for serum AMH concentration assessment is drawn. Blood serum is stored at -80C and AMH concentration assessment is performed in one badge.
4. Withdrawal of individual subjects Subjects can leave the study at any time for any reason if they wish to do so without any consequences. After withdrawal the individual subjects will be replaced.
5. Premature termination of the study In case of serious adverse events (like postoperative haemorrhage).

SAFETY REPORTING

1. In accordance to section 10, subsection 1, of the WMO, the investigator will inform the subjects and the reviewing accredited Medical Ethical Committee (METC) if anything occurs, on the basis of which it appears that the disadvantages of participation may be significantly greater than was foreseen in the research proposal. The study will be suspended pending further review by the accredited METC, except insofar as suspension would jeopardize the subjects' health. The investigator will take care that all subjects are kept informed.
2. Adverse and serious adverse events All Serious Adverse Event (SAE) s will be reported to the accredited METC that approved the protocol.

STATISTICAL ANALYSIS Data will both be described qualitatively and quantitatively. Student t-test will be applied to study differences in hormone levels between the groups.

ETHICAL CONSIDERATIONS

1. The study will be conducted according to the principles of the Declaration of Helsinki (2nd edition, 2009) and in accordance with the Medical Research Involving Human Subjects Act (WMO).
2. Patients will be recruited at the outpatient clinic when a decision is made for hysterectomy (abdominal or laparoscopic) on benign indication. They will receive oral information from their gynecologist and an information letter will be handed out (a telephone number will be stated which patients can call for extra information). On the day of preoperative admission (mostly one day preoperative) the gynecologist will answer any remaining questions and the informed consent will be signed by both the patient and the gynecologist. Patients on oral contraceptives will stop using these at least two weeks prior to the operation.
3. Literature on the effects of salpingectomy during hysterectomy for benign gynecological conditions on the ovarian reserve is very scant, but the one available study does not show any adverse effects. Furthermore, the chance of a postoperative hemorrhage is increased (estimated 1%). We believe that, in the light of the burden and risk, this study is justified since the prophylactic removal of the Fallopian tubes might diminish the risk of serous ovarian carcinomas (life time risk around 1%).

ADMINISTRATIVE ASPECTS AND PUBLICATION

1. Data will be collected from the participating hospitals by one study medical doctor. Together with the principal investigator (s)he has access to the source data which are coded by a case number. The key to the code is safeguarded in the safe from the TweeSteden hospital, Tilburg, The Netherlands. Data and human material will be kept for seven years (or fifteen with patient consent). Data security is assured by the fact that one medical doctor collects the data. The privacy of the participants is protected by the fact that the data is coded.
2. The investigator will submit a summary of the progress of the trial to the accredited METC once a year. Information will be provided on the date of inclusion of the first subject, numbers of subjects included and numbers of subjects that have completed the trial, serious adverse events / serious adverse reactions, other problems, and amendments.
3. The investigator will notify the accredited METC of the end of the study within a period of 8 weeks. The end of the study is defined as the last patient's last visit. In case the study is ended prematurely, the investigator will notify the accredited METC, including the reasons for the premature termination. Within one year after the end of the study, the investigator will submit a final study report with the results of the study, including any publications/abstracts of the study, to the accredited METC.
4. The data will be published in peer reviewed medical journals as well as presented in abstracts at medical conferences.

ELIGIBILITY:
Inclusion Criteria:

* hysterectomy (abdominally or laparoscopically) for benign indications
* premenopausal
* age >36 < 55

Exclusion Criteria:

* history of cancer
* hereditary cancer in the family
* previous intraluminal tubal occlusion
* previous salpingitis
* failure to perform a tubectomy during hysterectomy

Ages: 36 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Anti Mullerian Hormone | at baseline and on average six months after the operation
  Difference, if any, in concentration of Anti Mullerian Hormone one day prior to hysterectomy and on average around six months after surgery between the study groups (hysterectomy alone versus hysterectomy and tubectomy).

SECONDARY OUTCOMES:
Dysplasia | on average six months after the operation
  Analysis of the incidence of dysplastic lesions (defined as: nuclear atypia, pilling of epithelial cells, multiple mitosis), if any, in the removed Fallopian tubes by light microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen M Piek, MD. PhD., Principal Investigator — Gynaecologisch Oncologisch Centrum Zuid
Locations (5):
- Netherlands (5):
  - Radboudumc, Nijmegen, Gelderland
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch, North Brabant
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Elisabeth ziekenhuis, Tilburg, North Brabant
  - TweeStedenziekenhuis, Tilburg, North Brabant

REFERENCES:
- [Background] Piek JM, van Diest PJ, Zweemer RP, Kenemans P, Verheijen RH. Tubal ligation and risk of ovarian cancer. Lancet. 2001 Sep 8;358(9284):844. doi: 10.1016/S0140-6736(01)05992-X. No abstract available. PMID 11570411
- [Background] Kurman RJ, Shih IeM. The origin and pathogenesis of epithelial ovarian cancer: a proposed unifying theory. Am J Surg Pathol. 2010 Mar;34(3):433-43. doi: 10.1097/PAS.0b013e3181cf3d79. PMID 20154587
- [Background] Crum CP. Intercepting pelvic cancer in the distal fallopian tube: theories and realities. Mol Oncol. 2009 Apr;3(2):165-70. doi: 10.1016/j.molonc.2009.01.004. Epub 2009 Feb 3. PMID 19383378
- [Background] Sezik M, Ozkaya O, Demir F, Sezik HT, Kaya H. Total salpingectomy during abdominal hysterectomy: effects on ovarian reserve and ovarian stromal blood flow. J Obstet Gynaecol Res. 2007 Dec;33(6):863-9. doi: 10.1111/j.1447-0756.2007.00669.x. PMID 18001455
- [Background] Narod SA, Sun P, Ghadirian P, Lynch H, Isaacs C, Garber J, Weber B, Karlan B, Fishman D, Rosen B, Tung N, Neuhausen SL. Tubal ligation and risk of ovarian cancer in carriers of BRCA1 or BRCA2 mutations: a case-control study. Lancet. 2001 May 12;357(9267):1467-70. doi: 10.1016/s0140-6736(00)04642-0. PMID 11377596